CLINICAL TRIAL: NCT03447678
Title: Phase II Study to Test Pembrolizumab (MK-3475) in First Line Treatment of Advanced NSCLC Patients With PD-L1 Low Tumors (<50%)_ PEOPLE TRIAL (Pembrolizumab in Pd-L1 Low Expressors).
Brief Title: Pembrolizumab in First Line Treatment of Advanced NSCLC Patients With PD-L1 Low Tumors.
Acronym: PEOPLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 178-17
Record Dates: First submitted 2018-02-13; First posted 2018-02-27 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): subjects with PD-L1 low (PD-L1Lo), EGFR wt, EML4/ALK fusion negative NSCLC
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — humanized antibody used in cancer immunotherapy

SUMMARY:
This is a prospective, monocentric, open label, phase II trial of intravenous (IV) Pembrolizumab monotherapy in subjects previously untreated for their stage IIIB-IV, PD-L1 low non small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Approximately 65 subjects with PD-L1 low (PD-L1Lo), EGFR wt, EML4/ALK fusion negative NSCLC will be enrolled in this trial for examination of the biological characteristics associated to efficacy and safety of Pembrolizumab. Subjects will receive Pembrolizumab iv at dose of 200 mg every three weeks. Subjects will be evaluated every 9 weeks (63 +/- 3 days) with radiographic imaging to assess response to treatment. Subjects will continue with the assigned study treatment until RECIST-defined progression of disease, unacceptable toxicity or consent withdrawal.

Treatment with Pembrolizumab will continue until two years of therapy have been administered, documented disease progression, unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, or administrative reasons. Pembrolizumab treated subjects who obtain a confirmed Complete Response (CR) per RECIST 1.1 may consider stopping trial treatment. These subjects may be eligible for re-treatment with Pembrolizumab after they have experienced radiographic disease progression at the discretion of the investigator, this re-treatment will be the Second Course Phase.

ELIGIBILITY:
Inclusion Criteria:

1. Have a confirmed diagnosis of NSCLC in stage IIIB/ IV. Do not have an EGFR sensitizing (activating) mutation or ALK translocation and have a PD-L1 "low" (<50%) tumor as determined by immunohistochemistry with anti-PD-L1 antibody (DAKO 22C3). Have not received prior systemic chemotherapy treatment for advanced NSCLC. Subjects with non-squamous histologies will not be enrolled until the EGFR mutation status and/or ALK translocation status is available. For patients enrolled who are known to have a tumor of predominantly squamous histology, molecular testing for EGFR and ALK translocation will not be required .
2. Be willing and able to provide written informed consent/assent for the trial.
3. Be >=18 years of age on day of signing informed consent.
4. Have measurable disease based on RECIST 1.1.
5. Be willing to provide tissue from archived histological specimen or newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 45 days prior to initiation of treatment on Day 1.
6. Have a performance status of 0 or 1 on the ECOG Performance Scale.
7. Demonstrate adequate organ function
8. All screening labs should be performed within 10 days of treatment initiation
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
10. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
11. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
12. No history of active malignancy requiring treatment

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Has an EGFR sensitizing mutation and/or an ALK translocation.
2. Has a PD-L1 expression assessed as "high" by the central laboratory
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has a known history of active TB (Bacillus Tuberculosis).
5. Hypersensitivity to Pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subjects received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has a history of non-infectious pneumonitis that required steroids or has current pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Immune biomarkers | 3 years
  tumor infiltrating lymphocytes in patients whose tumors have a low PD_L1 expression
Immune biomarkers | 3 years
  infiltrating T cells that upregulate PD-1
Immune biomarkers | 3 years
  inhibitory receptors such as TIM-3, LAG-3 and TIGIT
Immune biomarkers | 3 years
  type of cells being positive for PD-L1(neoplastic cells vs infiltrating immune cells)
Immune biomarkers | 3 years
  presence and phenotype of tumor-infiltrating lymphocytes in the pre-therapy lesions of patients with low expression of PD-L1
Immune biomarkers | 3 years
  levels of CD3+, CD4+, CD8+ lymphocytes
Immune biomarkers | 3 years
  expression, in TIL, of markers of functional differentiation to cytolytic stage such as granzyme B and TIA-1, or maturation to memory stage (CD45RO)
Immune biomarkers | 3 years
  expression of PD1+ by TIL
Immune biomarkers | 3 years
  expression of PD-L1 on neoplastic cells vs immune cells
Immune biomarkers | 3 years
  expression of inhibitory receptors as LAG-3, TIM-3 and TIGIT
Immune biomarkers | 3 years
  frequency of FOXP3+ lymphocytes, as well as of CD11b+ CD33+ MDSCs, in pre-therapy lesions

SECONDARY OUTCOMES:
Immune biomarkers distribution between pre and post Pembrolizumab treatment | 3 years
  tumor infiltrating lymphocytes in patients whose tumors have a low PD_L1 expression
Immune biomarkers distribution between pre and post Pembrolizumab treatment | 3 years
  infiltrating T cells that upregulate PD-1
Immune biomarkers distribution between pre and post Pembrolizumab treatment | 3 years
  inhibitory receptors such as TIM-3, LAG-3 and TIGIT
Immune biomarkers distribution between pre and post Pembrolizumab treatment | 3 years
  type of cells being positive for PD-L1(neoplastic cells vs infiltrating immune cells)
Immune biomarkers distribution between pre and post Pembrolizumab treatment | 3 years
  presence and phenotype of tumor-infiltrating lymphocytes in the pre-therapy lesions of patients with low expression of PD-L1
Immune biomarkers distribution between pre and post Pembrolizumab treatment | 3 years
  levels of CD3+, CD4+, CD8+ lymphocytes
Immune biomarkers distribution between pre and post Pembrolizumab treatment | 3 years
  expression, in TIL, of markers of functional differentiation to cytolytic stage such as granzyme B and TIA-1, or maturation to memory stage (CD45RO)
Immune biomarkers distribution between pre and post Pembrolizumab treatment | 3 years
  expression of PD1+ by TIL
Immune biomarkers distribution between pre and post Pembrolizumab treatment | 3 years
  expression of PD-L1 on neoplastic cells vs immune cells
Immune biomarkers distribution between pre and post Pembrolizumab treatment | 3 years
  expression of inhibitory receptors as LAG-3, TIM-3 and TIGIT
Immune biomarkers distribution between pre and post Pembrolizumab treatment | 3 years
  frequency of FOXP3+ lymphocytes, as well as of CD11b+ CD33+ MDSCs, in pre-therapy lesions
Activity endpoints | from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease are objectively documented, assessed up to 3 years
  Response Duration (DoR)
Activity endpoints | 3 years
  Objective Response Rate (ORR)
Activity endpoints | 3 years
  Disease Control Rate (DCR)
Effectiveness of Pembrolizumab treatment | from the time of enrollment to death due to any reasons, assessed up to 3 years
  Overall Survival (OS) will be used as effectiveness endpoint
Safety of Pembrolizumab treatment. | 3 years
  Adverse events will be monitored throughout the trial and graded in severity according to the guidelines outlined in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4. A particular attention will be placed in the evaluation of potential Immune related adverse events (IrAE)
Patient Reported health status for physical, mental and social well-being | 3 years
  The patient Reported Outcomes Measurement Information System (PROMIS) provides measures of health status that assess physical, mental and social well-being from the patient prospective.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Chiara Garassino, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korman A, Chen B, Wang C, Wu L, Cardarelli P, Selby M. Activity of anti-PD-1 in murine tumor models: role of
- [Background] Rizvi NA,et al. Safety and clinical activity of Pembrolizumab as initial therapy in patients with advanced non-small cell lung cancer (NSCLC). Presented at the ASCO Meeting 2014. abstract 8007.
- [Background] Garon EB, et al. Safety and clinical activity of Pembrolizumab in previously treated patients (pts) with non-small cell lung cancer (NSCLC). Presented at the ASCO Meeting 2014. abstract 8020.
- [Background] Harriet M. Kluger, Sarah B. Goldberg, Mario Sznol, John Tsiouris, Alexander Vortmeyer, Lucia Jilaveanu, Amanda L. Ralabate, Angel L. Rivera, Matthew M. Burke, Upendra P. Hegbe, Justine Vanessa Cohen, Xiaopan Yao, Stephanie Speaker, Matthew Madura, Elizabeth Knapp-Perry, Amit Mahajan, Veronica Chiang. Safety and activity of Pembrolizumab in melanoma patients with untreated brain metastases. 2015 ASCO annual meeting
- [Background] A.S. Berghoff, C. Inan, G. Ricken, G. Widhalm, K. Dieckmann, P. Birner, F. Oberndorfer, B. Dome, R. Bartsch, C. Zielinski and M. Preusser. Tumor-infiltrating lymphocytes (tils) and pd-l1 expression in non- small cell lung cancer brain metastases (bm) and matched primary tumors (pt). Ann oncol (2014) 25 (suppl 4): iv465-iv466.
- [Result] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428
- [Result] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Result] Sharpe AH, Freeman GJ. The B7-CD28 superfamily. Nat Rev Immunol. 2002 Feb;2(2):116-26. doi: 10.1038/nri727. PMID 11910893
- [Result] Brown JA, Dorfman DM, Ma FR, Sullivan EL, Munoz O, Wood CR, Greenfield EA, Freeman GJ. Blockade of programmed death-1 ligands on dendritic cells enhances T cell activation and cytokine production. J Immunol. 2003 Feb 1;170(3):1257-66. doi: 10.4049/jimmunol.170.3.1257. PMID 12538684
- [Result] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Result] Thompson RH, Dong H, Lohse CM, Leibovich BC, Blute ML, Cheville JC, Kwon ED. PD-1 is expressed by tumor-infiltrating immune cells and is associated with poor outcome for patients with renal cell carcinoma. Clin Cancer Res. 2007 Mar 15;13(6):1757-61. doi: 10.1158/1078-0432.CCR-06-2599. PMID 17363529
- [Result] Hino R, Kabashima K, Kato Y, Yagi H, Nakamura M, Honjo T, Okazaki T, Tokura Y. Tumor cell expression of programmed cell death-1 ligand 1 is a prognostic factor for malignant melanoma. Cancer. 2010 Apr 1;116(7):1757-66. doi: 10.1002/cncr.24899. PMID 20143437
- [Result] Nomi T, Sho M, Akahori T, Hamada K, Kubo A, Kanehiro H, Nakamura S, Enomoto K, Yagita H, Azuma M, Nakajima Y. Clinical significance and therapeutic potential of the programmed death-1 ligand/programmed death-1 pathway in human pancreatic cancer. Clin Cancer Res. 2007 Apr 1;13(7):2151-7. doi: 10.1158/1078-0432.CCR-06-2746. PMID 17404099
- [Result] Gao Q, Wang XY, Qiu SJ, Yamato I, Sho M, Nakajima Y, Zhou J, Li BZ, Shi YH, Xiao YS, Xu Y, Fan J. Overexpression of PD-L1 significantly associates with tumor aggressiveness and postoperative recurrence in human hepatocellular carcinoma. Clin Cancer Res. 2009 Feb 1;15(3):971-9. doi: 10.1158/1078-0432.CCR-08-1608. PMID 19188168
- [Result] Hamanishi J, Mandai M, Iwasaki M, Okazaki T, Tanaka Y, Yamaguchi K, Higuchi T, Yagi H, Takakura K, Minato N, Honjo T, Fujii S. Programmed cell death 1 ligand 1 and tumor-infiltrating CD8+ T lymphocytes are prognostic factors of human ovarian cancer. Proc Natl Acad Sci U S A. 2007 Feb 27;104(9):3360-5. doi: 10.1073/pnas.0611533104. Epub 2007 Feb 21. PMID 17360651
- [Result] Fourcade J, Kudela P, Sun Z, Shen H, Land SR, Lenzner D, Guillaume P, Luescher IF, Sander C, Ferrone S, Kirkwood JM, Zarour HM. PD-1 is a regulator of NY-ESO-1-specific CD8+ T cell expansion in melanoma patients. J Immunol. 2009 May 1;182(9):5240-9. doi: 10.4049/jimmunol.0803245. PMID 19380770
- [Result] Cai G, Karni A, Oliveira EM, Weiner HL, Hafler DA, Freeman GJ. PD-1 ligands, negative regulators for activation of naive, memory, and recently activated human CD4+ T cells. Cell Immunol. 2004 Aug;230(2):89-98. doi: 10.1016/j.cellimm.2004.09.004. PMID 15598424
- [Result] Blank C, Mackensen A. Contribution of the PD-L1/PD-1 pathway to T-cell exhaustion: an update on implications for chronic infections and tumor evasion. Cancer Immunol Immunother. 2007 May;56(5):739-45. doi: 10.1007/s00262-006-0272-1. Epub 2006 Dec 29. PMID 17195077
- [Result] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Result] Tsushima F, Tanaka K, Otsuki N, Youngnak P, Iwai H, Omura K, Azuma M. Predominant expression of B7-H1 and its immunoregulatory roles in oral squamous cell carcinoma. Oral Oncol. 2006 Mar;42(3):268-74. doi: 10.1016/j.oraloncology.2005.07.013. Epub 2005 Nov 3. PMID 16271509
- [Result] Oble DA, Loewe R, Yu P, Mihm MC Jr. Focus on TILs: prognostic significance of tumor infiltrating lymphocytes in human melanoma. Cancer Immun. 2009 Apr 2;9:3. PMID 19338264
- [Result] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Result] Patnaik A, Kang SP, Rasco D, Papadopoulos KP, Elassaiss-Schaap J, Beeram M, Drengler R, Chen C, Smith L, Espino G, Gergich K, Delgado L, Daud A, Lindia JA, Li XN, Pierce RH, Yearley JH, Wu D, Laterza O, Lehnert M, Iannone R, Tolcher AW. Phase I Study of Pembrolizumab (MK-3475; Anti-PD-1 Monoclonal Antibody) in Patients with Advanced Solid Tumors. Clin Cancer Res. 2015 Oct 1;21(19):4286-93. doi: 10.1158/1078-0432.CCR-14-2607. Epub 2015 May 14. PMID 25977344
- [Result] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Result] Chapman PB, Hauschild A, Robert C, Haanen JB, Ascierto P, Larkin J, Dummer R, Garbe C, Testori A, Maio M, Hogg D, Lorigan P, Lebbe C, Jouary T, Schadendorf D, Ribas A, O'Day SJ, Sosman JA, Kirkwood JM, Eggermont AM, Dreno B, Nolop K, Li J, Nelson B, Hou J, Lee RJ, Flaherty KT, McArthur GA; BRIM-3 Study Group. Improved survival with vemurafenib in melanoma with BRAF V600E mutation. N Engl J Med. 2011 Jun 30;364(26):2507-16. doi: 10.1056/NEJMoa1103782. Epub 2011 Jun 5. PMID 21639808
- [Result] Robert C, Thomas L, Bondarenko I, O'Day S, Weber J, Garbe C, Lebbe C, Baurain JF, Testori A, Grob JJ, Davidson N, Richards J, Maio M, Hauschild A, Miller WH Jr, Gascon P, Lotem M, Harmankaya K, Ibrahim R, Francis S, Chen TT, Humphrey R, Hoos A, Wolchok JD. Ipilimumab plus dacarbazine for previously untreated metastatic melanoma. N Engl J Med. 2011 Jun 30;364(26):2517-26. doi: 10.1056/NEJMoa1104621. Epub 2011 Jun 5. PMID 21639810
- [Result] Bellati F, Visconti V, Napoletano C, Antonilli M, Frati L, Panici PB, Nuti M. Immunology of gynecologic neoplasms: analysis of the prognostic significance of the immune status. Curr Cancer Drug Targets. 2009 Jun;9(4):541-65. doi: 10.2174/156800909788486722. PMID 19519321
- [Result] Ruffell B, DeNardo DG, Affara NI, Coussens LM. Lymphocytes in cancer development: polarization towards pro-tumor immunity. Cytokine Growth Factor Rev. 2010 Feb;21(1):3-10. doi: 10.1016/j.cytogfr.2009.11.002. Epub 2009 Dec 11. PMID 20005150
- [Result] Shirabe K, Motomura T, Muto J, Toshima T, Matono R, Mano Y, Takeishi K, Ijichi H, Harada N, Uchiyama H, Yoshizumi T, Taketomi A, Maehara Y. Tumor-infiltrating lymphocytes and hepatocellular carcinoma: pathology and clinical management. Int J Clin Oncol. 2010 Dec;15(6):552-8. doi: 10.1007/s10147-010-0131-0. Epub 2010 Oct 21. PMID 20963618
- [Result] Al-Shibli K, Al-Saad S, Andersen S, Donnem T, Bremnes RM, Busund LT. The prognostic value of intraepithelial and stromal CD3-, CD117- and CD138-positive cells in non-small cell lung carcinoma. APMIS. 2010 May;118(5):371-82. doi: 10.1111/j.1600-0463.2010.02609.x. PMID 20477813
- [Result] Clark CE, Beatty GL, Vonderheide RH. Immunosurveillance of pancreatic adenocarcinoma: insights from genetically engineered mouse models of cancer. Cancer Lett. 2009 Jun 28;279(1):1-7. doi: 10.1016/j.canlet.2008.09.037. Epub 2008 Nov 14. PMID 19013709
- [Result] Diederichsen AC, Hjelmborg Jv, Christensen PB, Zeuthen J, Fenger C. Prognostic value of the CD4+/CD8+ ratio of tumour infiltrating lymphocytes in colorectal cancer and HLA-DR expression on tumour cells. Cancer Immunol Immunother. 2003 Jul;52(7):423-8. doi: 10.1007/s00262-003-0388-5. Epub 2003 Apr 15. PMID 12695859
- [Result] Gao Q, Qiu SJ, Fan J, Zhou J, Wang XY, Xiao YS, Xu Y, Li YW, Tang ZY. Intratumoral balance of regulatory and cytotoxic T cells is associated with prognosis of hepatocellular carcinoma after resection. J Clin Oncol. 2007 Jun 20;25(18):2586-93. doi: 10.1200/JCO.2006.09.4565. PMID 17577038
- [Result] Hillen F, Baeten CI, van de Winkel A, Creytens D, van der Schaft DW, Winnepenninckx V, Griffioen AW. Leukocyte infiltration and tumor cell plasticity are parameters of aggressiveness in primary cutaneous melanoma. Cancer Immunol Immunother. 2008 Jan;57(1):97-106. doi: 10.1007/s00262-007-0353-9. Epub 2007 Jun 30. PMID 17602225
- [Result] Laghi L, Bianchi P, Miranda E, Balladore E, Pacetti V, Grizzi F, Allavena P, Torri V, Repici A, Santoro A, Mantovani A, Roncalli M, Malesci A. CD3+ cells at the invasive margin of deeply invading (pT3-T4) colorectal cancer and risk of post-surgical metastasis: a longitudinal study. Lancet Oncol. 2009 Sep;10(9):877-84. doi: 10.1016/S1470-2045(09)70186-X. Epub 2009 Aug 3. PMID 19656725
- [Result] Li JF, Chu YW, Wang GM, Zhu TY, Rong RM, Hou J, Xu M. The prognostic value of peritumoral regulatory T cells and its correlation with intratumoral cyclooxygenase-2 expression in clear cell renal cell carcinoma. BJU Int. 2009 Feb;103(3):399-405. doi: 10.1111/j.1464-410X.2008.08151.x. Epub 2008 Nov 19. PMID 19021626
- [Result] Nemolato S, Fanni D, Naccarato AG, Ravarino A, Bevilacqua G, Faa G. Lymphoepitelioma-like hepatocellular carcinoma: a case report and a review of the literature. World J Gastroenterol. 2008 Aug 7;14(29):4694-6. doi: 10.3748/wjg.14.4694. PMID 18698686
- [Result] Nobili C, Degrate L, Caprotti R, Franciosi C, Leone BE, Trezzi R, Romano F, Uggeri F, Uggeri F. Prolonged survival of a patient affected by pancreatic adenocarcinoma with massive lymphocyte and dendritic cell infiltration after interleukin-2 immunotherapy. Report of a case. Tumori. 2008 May-Jun;94(3):426-30. doi: 10.1177/030089160809400323. PMID 18705415
- [Result] Oshikiri T, Miyamoto M, Shichinohe T, Suzuoki M, Hiraoka K, Nakakubo Y, Shinohara T, Itoh T, Kondo S, Katoh H. Prognostic value of intratumoral CD8+ T lymphocyte in extrahepatic bile duct carcinoma as essential immune response. J Surg Oncol. 2003 Dec;84(4):224-8. doi: 10.1002/jso.10321. PMID 14756433
- [Result] Piersma SJ, Welters MJ, van der Burg SH. Tumor-specific regulatory T cells in cancer patients. Hum Immunol. 2008 Apr-May;69(4-5):241-9. doi: 10.1016/j.humimm.2008.02.005. Epub 2008 Mar 28. PMID 18486758
- [Result] Rao UN, Lee SJ, Luo W, Mihm MC Jr, Kirkwood JM. Presence of tumor-infiltrating lymphocytes and a dominant nodule within primary melanoma are prognostic factors for relapse-free survival of patients with thick (t4) primary melanoma: pathologic analysis of the e1690 and e1694 intergroup trials. Am J Clin Pathol. 2010 Apr;133(4):646-53. doi: 10.1309/AJCPTXMEFOVYWDA6. PMID 20231618
- [Result] Sasaki A, Tanaka F, Mimori K, Inoue H, Kai S, Shibata K, Ohta M, Kitano S, Mori M. Prognostic value of tumor-infiltrating FOXP3+ regulatory T cells in patients with hepatocellular carcinoma. Eur J Surg Oncol. 2008 Feb;34(2):173-9. doi: 10.1016/j.ejso.2007.08.008. Epub 2007 Oct 10. PMID 17928188
- [Result] Shen Z, Zhou S, Wang Y, Li RL, Zhong C, Liang C, Sun Y. Higher intratumoral infiltrated Foxp3+ Treg numbers and Foxp3+/CD8+ ratio are associated with adverse prognosis in resectable gastric cancer. J Cancer Res Clin Oncol. 2010 Oct;136(10):1585-95. doi: 10.1007/s00432-010-0816-9. Epub 2010 Mar 11. PMID 20221835
- [Result] Talmadge JE, Donkor M, Scholar E. Inflammatory cell infiltration of tumors: Jekyll or Hyde. Cancer Metastasis Rev. 2007 Dec;26(3-4):373-400. doi: 10.1007/s10555-007-9072-0. PMID 17717638
- [Result] Usubutun A, Ayhan A, Uygur MC, Ozen H, Toklu C, Ruacan S. Prognostic factors in renal cell carcinoma. J Exp Clin Cancer Res. 1998 Mar;17(1):77-81. PMID 9646237
- [Result] Hiraoka N. Tumor-infiltrating lymphocytes and hepatocellular carcinoma: molecular biology. Int J Clin Oncol. 2010 Dec;15(6):544-51. doi: 10.1007/s10147-010-0130-1. Epub 2010 Oct 6. PMID 20924634
- [Result] Hodi FS, Dranoff G. The biologic importance of tumor-infiltrating lymphocytes. J Cutan Pathol. 2010 Apr;37 Suppl 1(0 1):48-53. doi: 10.1111/j.1600-0560.2010.01506.x. PMID 20482675
- [Result] Kloor M. Lymphocyte infiltration and prognosis in colorectal cancer. Lancet Oncol. 2009 Sep;10(9):840-1. doi: 10.1016/S1470-2045(09)70245-1. No abstract available. PMID 19717085
- [Result] Lee HE, Chae SW, Lee YJ, Kim MA, Lee HS, Lee BL, Kim WH. Prognostic implications of type and density of tumour-infiltrating lymphocytes in gastric cancer. Br J Cancer. 2008 Nov 18;99(10):1704-11. doi: 10.1038/sj.bjc.6604738. Epub 2008 Oct 21. PMID 18941457
- [Result] Leffers N, Gooden MJ, de Jong RA, Hoogeboom BN, ten Hoor KA, Hollema H, Boezen HM, van der Zee AG, Daemen T, Nijman HW. Prognostic significance of tumor-infiltrating T-lymphocytes in primary and metastatic lesions of advanced stage ovarian cancer. Cancer Immunol Immunother. 2009 Mar;58(3):449-59. doi: 10.1007/s00262-008-0583-5. Epub 2008 Sep 13. PMID 18791714
- [Result] Nishimura H, Honjo T, Minato N. Facilitation of beta selection and modification of positive selection in the thymus of PD-1-deficient mice. J Exp Med. 2000 Mar 6;191(5):891-8. doi: 10.1084/jem.191.5.891. PMID 10704469
- [Result] Polcher M, Braun M, Friedrichs N, Rudlowski C, Bercht E, Fimmers R, Sauerwald A, Keyver-Paik MD, Kubler K, Buttner R, Kuhn WC, Hernando JJ. Foxp3(+) cell infiltration and granzyme B(+)/Foxp3(+) cell ratio are associated with outcome in neoadjuvant chemotherapy-treated ovarian carcinoma. Cancer Immunol Immunother. 2010 Jun;59(6):909-19. doi: 10.1007/s00262-010-0817-1. Epub 2010 Jan 20. PMID 20087581
- [Result] Suzuki H, Chikazawa N, Tasaka T, Wada J, Yamasaki A, Kitaura Y, Sozaki M, Tanaka M, Onishi H, Morisaki T, Katano M. Intratumoral CD8(+) T/FOXP3 (+) cell ratio is a predictive marker for survival in patients with colorectal cancer. Cancer Immunol Immunother. 2010 May;59(5):653-61. doi: 10.1007/s00262-009-0781-9. Epub 2009 Nov 12. PMID 19908042
- [Result] Chew V, Tow C, Teo M, Wong HL, Chan J, Gehring A, Loh M, Bolze A, Quek R, Lee VK, Lee KH, Abastado JP, Toh HC, Nardin A. Inflammatory tumour microenvironment is associated with superior survival in hepatocellular carcinoma patients. J Hepatol. 2010 Mar;52(3):370-9. doi: 10.1016/j.jhep.2009.07.013. Epub 2009 Aug 3. PMID 19720422
- [Result] Liotta F, Gacci M, Frosali F, Querci V, Vittori G, Lapini A, Santarlasci V, Serni S, Cosmi L, Maggi L, Angeli R, Mazzinghi B, Romagnani P, Maggi E, Carini M, Romagnani S, Annunziato F. Frequency of regulatory T cells in peripheral blood and in tumour-infiltrating lymphocytes correlates with poor prognosis in renal cell carcinoma. BJU Int. 2011 May;107(9):1500-6. doi: 10.1111/j.1464-410X.2010.09555.x. Epub 2010 Aug 24. PMID 20735382
- [Result] Ropponen KM, Eskelinen MJ, Lipponen PK, Alhava E, Kosma VM. Prognostic value of tumour-infiltrating lymphocytes (TILs) in colorectal cancer. J Pathol. 1997 Jul;182(3):318-24. doi: 10.1002/(SICI)1096-9896(199707)182:33.0.CO;2-6. PMID 9349235
- [Result] Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, Royal RE, Kammula U, White DE, Mavroukakis SA, Rogers LJ, Gracia GJ, Jones SA, Mangiameli DP, Pelletier MM, Gea-Banacloche J, Robinson MR, Berman DM, Filie AC, Abati A, Rosenberg SA. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol. 2005 Apr 1;23(10):2346-57. doi: 10.1200/JCO.2005.00.240. PMID 15800326
- [Result] Hunder NN, Wallen H, Cao J, Hendricks DW, Reilly JZ, Rodmyre R, Jungbluth A, Gnjatic S, Thompson JA, Yee C. Treatment of metastatic melanoma with autologous CD4+ T cells against NY-ESO-1. N Engl J Med. 2008 Jun 19;358(25):2698-703. doi: 10.1056/NEJMoa0800251. PMID 18565862
- [Result] Okazaki T, Maeda A, Nishimura H, Kurosaki T, Honjo T. PD-1 immunoreceptor inhibits B cell receptor-mediated signaling by recruiting src homology 2-domain-containing tyrosine phosphatase 2 to phosphotyrosine. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):13866-71. doi: 10.1073/pnas.231486598. Epub 2001 Nov 6. PMID 11698646
- [Result] Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol. 2005;23:515-48. doi: 10.1146/annurev.immunol.23.021704.115611. PMID 15771580
- [Result] Hamid O, Robert C, Daud A, Hodi FS, Hwu WJ, Kefford R, Wolchok JD, Hersey P, Joseph RW, Weber JS, Dronca R, Gangadhar TC, Patnaik A, Zarour H, Joshua AM, Gergich K, Elassaiss-Schaap J, Algazi A, Mateus C, Boasberg P, Tumeh PC, Chmielowski B, Ebbinghaus SW, Li XN, Kang SP, Ribas A. Safety and tumor responses with lambrolizumab (anti-PD-1) in melanoma. N Engl J Med. 2013 Jul 11;369(2):134-44. doi: 10.1056/NEJMoa1305133. Epub 2013 Jun 2. PMID 23724846
- [Result] Peters S, Adjei AA, Gridelli C, Reck M, Kerr K, Felip E; ESMO Guidelines Working Group. Metastatic non-small-cell lung cancer (NSCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2012 Oct;23 Suppl 7:vii56-64. doi: 10.1093/annonc/mds226. No abstract available. PMID 22997455
- [Result] Scagliotti GV, Parikh P, von Pawel J, Biesma B, Vansteenkiste J, Manegold C, Serwatowski P, Gatzemeier U, Digumarti R, Zukin M, Lee JS, Mellemgaard A, Park K, Patil S, Rolski J, Goksel T, de Marinis F, Simms L, Sugarman KP, Gandara D. Phase III study comparing cisplatin plus gemcitabine with cisplatin plus pemetrexed in chemotherapy-naive patients with advanced-stage non-small-cell lung cancer. J Clin Oncol. 2008 Jul 20;26(21):3543-51. doi: 10.1200/JCO.2007.15.0375. Epub 2008 May 27. PMID 18506025
- [Result] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Result] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Result] Reck M, von Pawel J, Zatloukal P, Ramlau R, Gorbounova V, Hirsh V, Leighl N, Mezger J, Archer V, Moore N, Manegold C. Phase III trial of cisplatin plus gemcitabine with either placebo or bevacizumab as first-line therapy for nonsquamous non-small-cell lung cancer: AVAil. J Clin Oncol. 2009 Mar 10;27(8):1227-34. doi: 10.1200/JCO.2007.14.5466. Epub 2009 Feb 2. PMID 19188680
- [Result] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137
- [Result] Nishie K, Kawaguchi T, Tamiya A, Mimori T, Takeuchi N, Matsuda Y, Omachi N, Asami K, Okishio K, Atagi S, Okuma T, Kubo A, Maruyama Y, Kudoh S, Takada M. Epidermal growth factor receptor tyrosine kinase inhibitors beyond progressive disease: a retrospective analysis for Japanese patients with activating EGFR mutations. J Thorac Oncol. 2012 Nov;7(11):1722-7. doi: 10.1097/JTO.0b013e31826913f7. PMID 23059777
- [Result] Camidge DR, Bang YJ, Kwak EL, Iafrate AJ, Varella-Garcia M, Fox SB, Riely GJ, Solomon B, Ou SH, Kim DW, Salgia R, Fidias P, Engelman JA, Gandhi L, Janne PA, Costa DB, Shapiro GI, Lorusso P, Ruffner K, Stephenson P, Tang Y, Wilner K, Clark JW, Shaw AT. Activity and safety of crizotinib in patients with ALK-positive non-small-cell lung cancer: updated results from a phase 1 study. Lancet Oncol. 2012 Oct;13(10):1011-9. doi: 10.1016/S1470-2045(12)70344-3. Epub 2012 Sep 4. PMID 22954507
- [Result] Fukuoka M, Wu YL, Thongprasert S, Sunpaweravong P, Leong SS, Sriuranpong V, Chao TY, Nakagawa K, Chu DT, Saijo N, Duffield EL, Rukazenkov Y, Speake G, Jiang H, Armour AA, To KF, Yang JC, Mok TS. Biomarker analyses and final overall survival results from a phase III, randomized, open-label, first-line study of gefitinib versus carboplatin/paclitaxel in clinically selected patients with advanced non-small-cell lung cancer in Asia (IPASS). J Clin Oncol. 2011 Jul 20;29(21):2866-74. doi: 10.1200/JCO.2010.33.4235. Epub 2011 Jun 13. PMID 21670455
- [Result] Akbay EA, Koyama S, Carretero J, Altabef A, Tchaicha JH, Christensen CL, Mikse OR, Cherniack AD, Beauchamp EM, Pugh TJ, Wilkerson MD, Fecci PE, Butaney M, Reibel JB, Soucheray M, Cohoon TJ, Janne PA, Meyerson M, Hayes DN, Shapiro GI, Shimamura T, Sholl LM, Rodig SJ, Freeman GJ, Hammerman PS, Dranoff G, Wong KK. Activation of the PD-1 pathway contributes to immune escape in EGFR-driven lung tumors. Cancer Discov. 2013 Dec;3(12):1355-63. doi: 10.1158/2159-8290.CD-13-0310. Epub 2013 Sep 27. PMID 24078774
- [Result] Gettinger S, Herbst RS. B7-H1/PD-1 blockade therapy in non-small cell lung cancer: current status and future direction. Cancer J. 2014 Jul-Aug;20(4):281-9. doi: 10.1097/PPO.0000000000000063. PMID 25098289
- [Result] Velcheti V, Schalper KA, Carvajal DE, Anagnostou VK, Syrigos KN, Sznol M, Herbst RS, Gettinger SN, Chen L, Rimm DL. Programmed death ligand-1 expression in non-small cell lung cancer. Lab Invest. 2014 Jan;94(1):107-16. doi: 10.1038/labinvest.2013.130. Epub 2013 Nov 11. PMID 24217091
- [Result] Taube JM, Klein A, Brahmer JR, Xu H, Pan X, Kim JH, Chen L, Pardoll DM, Topalian SL, Anders RA. Association of PD-1, PD-1 ligands, and other features of the tumor immune microenvironment with response to anti-PD-1 therapy. Clin Cancer Res. 2014 Oct 1;20(19):5064-74. doi: 10.1158/1078-0432.CCR-13-3271. Epub 2014 Apr 8. PMID 24714771
- [Result] Bauer CA, Kim EY, Marangoni F, Carrizosa E, Claudio NM, Mempel TR. Dynamic Treg interactions with intratumoral APCs promote local CTL dysfunction. J Clin Invest. 2014 Jun;124(6):2425-40. doi: 10.1172/JCI66375. Epub 2014 May 8. PMID 24812664
- [Result] Highfill SL, Cui Y, Giles AJ, Smith JP, Zhang H, Morse E, Kaplan RN, Mackall CL. Disruption of CXCR2-mediated MDSC tumor trafficking enhances anti-PD1 efficacy. Sci Transl Med. 2014 May 21;6(237):237ra67. doi: 10.1126/scitranslmed.3007974. PMID 24848257
- [Result] Ascierto PA, Kalos M, Schaer DA, Callahan MK, Wolchok JD. Biomarkers for immunostimulatory monoclonal antibodies in combination strategies for melanoma and other tumor types. Clin Cancer Res. 2013 Mar 1;19(5):1009-20. doi: 10.1158/1078-0432.CCR-12-2982. PMID 23460532
- [Result] Ng Tang D, Shen Y, Sun J, Wen S, Wolchok JD, Yuan J, Allison JP, Sharma P. Increased frequency of ICOS+ CD4 T cells as a pharmacodynamic biomarker for anti-CTLA-4 therapy. Cancer Immunol Res. 2013 Oct;1(4):229-34. doi: 10.1158/2326-6066.CIR-13-0020. Epub 2013 Jul 31. PMID 24777852
- [Result] Pico de Coana Y, Poschke I, Gentilcore G, Mao Y, Nystrom M, Hansson J, Masucci GV, Kiessling R. Ipilimumab treatment results in an early decrease in the frequency of circulating granulocytic myeloid-derived suppressor cells as well as their Arginase1 production. Cancer Immunol Res. 2013 Sep;1(3):158-62. doi: 10.1158/2326-6066.CIR-13-0016. Epub 2013 Aug 2. PMID 24777678
- [Result] Tarhini AA, Edington H, Butterfield LH, Lin Y, Shuai Y, Tawbi H, Sander C, Yin Y, Holtzman M, Johnson J, Rao UN, Kirkwood JM. Immune monitoring of the circulation and the tumor microenvironment in patients with regionally advanced melanoma receiving neoadjuvant ipilimumab. PLoS One. 2014 Feb 3;9(2):e87705. doi: 10.1371/journal.pone.0087705. eCollection 2014. PMID 24498358
- [Result] Improta G, Pelosi G, Tamborini E, Donia M, Santinami M, de Braud F, Fraggetta F. Biological insights into BRAFV600 mutations in melanoma patient: Not mere therapeutic targets. Oncoimmunology. 2013 Aug 1;2(8):e25594. doi: 10.4161/onci.25594. Epub 2013 Jul 3. PMID 24179707
- [Result] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Result] Bellmunt J, de Wit R, Vaughn DJ, Fradet Y, Lee JL, Fong L, Vogelzang NJ, Climent MA, Petrylak DP, Choueiri TK, Necchi A, Gerritsen W, Gurney H, Quinn DI, Culine S, Sternberg CN, Mai Y, Poehlein CH, Perini RF, Bajorin DF; KEYNOTE-045 Investigators. Pembrolizumab as Second-Line Therapy for Advanced Urothelial Carcinoma. N Engl J Med. 2017 Mar 16;376(11):1015-1026. doi: 10.1056/NEJMoa1613683. Epub 2017 Feb 17. PMID 28212060
- [Result] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Result] Nghiem PT, Bhatia S, Lipson EJ, Kudchadkar RR, Miller NJ, Annamalai L, Berry S, Chartash EK, Daud A, Fling SP, Friedlander PA, Kluger HM, Kohrt HE, Lundgren L, Margolin K, Mitchell A, Olencki T, Pardoll DM, Reddy SA, Shantha EM, Sharfman WH, Sharon E, Shemanski LR, Shinohara MM, Sunshine JC, Taube JM, Thompson JA, Townson SM, Yearley JH, Topalian SL, Cheever MA. PD-1 Blockade with Pembrolizumab in Advanced Merkel-Cell Carcinoma. N Engl J Med. 2016 Jun 30;374(26):2542-52. doi: 10.1056/NEJMoa1603702. Epub 2016 Apr 19. PMID 27093365
- [Result] Garon EB, Rizvi NA, Hui R, Leighl N, Balmanoukian AS, Eder JP, Patnaik A, Aggarwal C, Gubens M, Horn L, Carcereny E, Ahn MJ, Felip E, Lee JS, Hellmann MD, Hamid O, Goldman JW, Soria JC, Dolled-Filhart M, Rutledge RZ, Zhang J, Lunceford JK, Rangwala R, Lubiniecki GM, Roach C, Emancipator K, Gandhi L; KEYNOTE-001 Investigators. Pembrolizumab for the treatment of non-small-cell lung cancer. N Engl J Med. 2015 May 21;372(21):2018-28. doi: 10.1056/NEJMoa1501824. Epub 2015 Apr 19. PMID 25891174
- [Result] Robert C, Schachter J, Long GV, Arance A, Grob JJ, Mortier L, Daud A, Carlino MS, McNeil C, Lotem M, Larkin J, Lorigan P, Neyns B, Blank CU, Hamid O, Mateus C, Shapira-Frommer R, Kosh M, Zhou H, Ibrahim N, Ebbinghaus S, Ribas A; KEYNOTE-006 investigators. Pembrolizumab versus Ipilimumab in Advanced Melanoma. N Engl J Med. 2015 Jun 25;372(26):2521-32. doi: 10.1056/NEJMoa1503093. Epub 2015 Apr 19. PMID 25891173
- [Result] Alley EW, Lopez J, Santoro A, Morosky A, Saraf S, Piperdi B, van Brummelen E. Clinical safety and activity of pembrolizumab in patients with malignant pleural mesothelioma (KEYNOTE-028): preliminary results from a non-randomised, open-label, phase 1b trial. Lancet Oncol. 2017 May;18(5):623-630. doi: 10.1016/S1470-2045(17)30169-9. Epub 2017 Mar 11. PMID 28291584
- [Result] Seiwert TY, Burtness B, Mehra R, Weiss J, Berger R, Eder JP, Heath K, McClanahan T, Lunceford J, Gause C, Cheng JD, Chow LQ. Safety and clinical activity of pembrolizumab for treatment of recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-012): an open-label, multicentre, phase 1b trial. Lancet Oncol. 2016 Jul;17(7):956-965. doi: 10.1016/S1470-2045(16)30066-3. Epub 2016 May 27. PMID 27247226
- [Result] Herbst RS, Baas P, Kim DW, Felip E, Perez-Gracia JL, Han JY, Molina J, Kim JH, Arvis CD, Ahn MJ, Majem M, Fidler MJ, de Castro G Jr, Garrido M, Lubiniecki GM, Shentu Y, Im E, Dolled-Filhart M, Garon EB. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small-cell lung cancer (KEYNOTE-010): a randomised controlled trial. Lancet. 2016 Apr 9;387(10027):1540-1550. doi: 10.1016/S0140-6736(15)01281-7. Epub 2015 Dec 19. PMID 26712084
- [Result] Ribas A, Puzanov I, Dummer R, Schadendorf D, Hamid O, Robert C, Hodi FS, Schachter J, Pavlick AC, Lewis KD, Cranmer LD, Blank CU, O'Day SJ, Ascierto PA, Salama AK, Margolin KA, Loquai C, Eigentler TK, Gangadhar TC, Carlino MS, Agarwala SS, Moschos SJ, Sosman JA, Goldinger SM, Shapira-Frommer R, Gonzalez R, Kirkwood JM, Wolchok JD, Eggermont A, Li XN, Zhou W, Zernhelt AM, Lis J, Ebbinghaus S, Kang SP, Daud A. Pembrolizumab versus investigator-choice chemotherapy for ipilimumab-refractory melanoma (KEYNOTE-002): a randomised, controlled, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):908-18. doi: 10.1016/S1470-2045(15)00083-2. Epub 2015 Jun 23. PMID 26115796
- [Result] Chow LQM, Haddad R, Gupta S, Mahipal A, Mehra R, Tahara M, Berger R, Eder JP, Burtness B, Lee SH, Keam B, Kang H, Muro K, Weiss J, Geva R, Lin CC, Chung HC, Meister A, Dolled-Filhart M, Pathiraja K, Cheng JD, Seiwert TY. Antitumor Activity of Pembrolizumab in Biomarker-Unselected Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma: Results From the Phase Ib KEYNOTE-012 Expansion Cohort. J Clin Oncol. 2016 Nov 10;34(32):3838-3845. doi: 10.1200/JCO.2016.68.1478. Epub 2016 Sep 30. PMID 27646946
- [Result] Daud AI, Wolchok JD, Robert C, Hwu WJ, Weber JS, Ribas A, Hodi FS, Joshua AM, Kefford R, Hersey P, Joseph R, Gangadhar TC, Dronca R, Patnaik A, Zarour H, Roach C, Toland G, Lunceford JK, Li XN, Emancipator K, Dolled-Filhart M, Kang SP, Ebbinghaus S, Hamid O. Programmed Death-Ligand 1 Expression and Response to the Anti-Programmed Death 1 Antibody Pembrolizumab in Melanoma. J Clin Oncol. 2016 Dec;34(34):4102-4109. doi: 10.1200/JCO.2016.67.2477. Epub 2016 Oct 31. PMID 27863197